CLINICAL TRIAL: NCT02393989
Title: Three-Year Clinical Evaluation of Bonded Posterior Restorations: Amalgam vs Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Hande Kemaloglu, Dr, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-3/50
Record Dates: First submitted 2015-03-10; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Class II Lesions

ARMS (1):
- Active comparator (Experimental): posterior restorations
  Interventions: Procedure: posterior restoration

INTERVENTIONS:
Procedure: posterior restoration — restorations for caries effected teeth

SUMMARY:
Background: This 3-year clinical trial compared the performance and post-operative sensitivity of a posterior resin composite with that of bonded-amalgam in large sized cavities. Additionally, it was evaluated whether resin composite could be an alternative for bonded amalgam.

Methods: This was a randomized clinical trial. Patients in need of at least two posterior restorations were recruited. Authors randomly assigned one half of the restorations to receive bonded-amalgam and the other half to composite restorations. Forty bonded-amalgams and composites were evaluated for their performance on modified Ryge criteria and post-operative sensitivity using VAS for 36-months.

ELIGIBILITY:
Inclusion Criteria:

To be included, the teeth to be restored had to:

1. be asymptomatic
2. have occlusal and adjacent teeth in contact
3. have cavity sizes exceeding the one-third of the bucco-lingual distance between cusp tips -

Exclusion Criteria:

* Patients with periodontitis, poor oral hygiene, bruxism or a history of allergic reactions to any of the materials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Modified Ryge Criteria | 3 years